CLINICAL TRIAL: NCT01498692
Title: PLATINUM: A Prospective, Randomized, Multicenter Trial to Assess an Everolimus-Eluting Coronary Stent System (PROMUS Element™) for the Treatment of up to Two De Novo Coronary Artery Lesions - Small Vessel Sub-trial
Brief Title: The PLATINUM Clinical Trial to Assess the PROMUS Element Stent System for Treatment of De Novo Coronary Artery Lesions in Small Vessels
Acronym: PLATINUM SV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2046A
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Results first posted 2012-02-13 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Disease
Keywords: drug-eluting stents; DES; atherosclerotic
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PROMUS Element (Experimental): Patients enrolled in the study to receive treatment with the PROMUS Element everolimus-eluting stent
  Interventions: Device: PROMUS Element Coronary Stent System

INTERVENTIONS:
Device: PROMUS Element Coronary Stent System — PROMUS Element is a device/drug combination product composed of two components, a device (coronary stent system including a platinum chromium stent platform) and a drug product (a formulation of everolimus contained in a polymer coating)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the PROMUS Element™ Everolimus-Eluting Coronary Stent System for the treatment of patients with up to 2 de novo atherosclerotic coronary artery lesions. The lesions can be located in vessels that are smaller than average-sized.

DETAILED DESCRIPTION:
The wide-spread use of drug-eluting stents (DES) has evolved as standard of care in de novo lesions. The proposed study will evaluate the safety and effectiveness of PROMUS Element for the treatment of de novo atherosclerotic lesions in native coronary arteries. The study design is consistent with the draft guidance for industry titled, "Coronary Drug-Eluting Stents - Nonclinical and Clinical Studies" (March 2008).

During the trial, thienopyridines must be administered according to the 2007 American College of Cardiology (ACC)/American Heart Association (AHA)/Society for Cardiovascular Angiography and Interventions (SCAI) guidelines, which recommended that clopidogrel (75 mg daily) or ticlopidine (250 mg twice daily) be prescribed after stent implantation for at least 6 months in all patients, and for at least 12 months in patients who are not at high risk of bleeding. For sites in the United States, the use of prasugrel is not allowed as part of the PLATINUM Clinical Trial. For sites in other countries, prasugrel may be prescribed according to its approved dosing in countries in which it is available. For patients taking aspirin daily a loading dose is recommended; for patients who have not been taking aspirin daily, aspirin must be administered as a loading dose. Patients continue to take aspirin indefinitely to reduce the risk of thrombosis.

This PLATINUM Small Vessel study is a sub-trial associated with the PLATINUM Workhorse Randomized Controlled Trial, which is registered under NCT00823212.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age
* Patient (or legal guardian) understands study requirements and treatment procedures and provides written informed consent before any study-specific tests or procedures are performed
* For patients less than 20 years of age enrolled at a Japanese site, patient and patient's legal representative must provide written informed consent before any study-specific tests or procedures are performed
* Patient is eligible for percutaneous coronary intervention (PCI)
* Patient has documented stable angina pectoris or documented silent ischemia; or unstable angina pectoris
* Patient is an acceptable candidate for coronary artery bypass grafting (CABG)
* Patient has a left ventricular ejection fraction (LVEF) >=30% as measured within 30 days prior to enrollment
* Patient is willing to comply with all protocol-required follow-up evaluations

Angiographic Inclusion Criteria (visual estimate):

- Target lesion must be a de novo lesion located in a native coronary artery with a visually estimated reference vessel diameter ≥2.25 mm and <2.5 mm. Target lesion length must measure ≤28 mm by visual estimate. Target lesion must be located in a major coronary artery or branch with visually estimated stenosis ≥50% and <100% with Thrombolysis In Myocardial Infarction (TIMI) flow >1.

Exclusion Criteria:

* Patient has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute myocardial infarction (MI)
* Patient has had a known diagnosis of recent MI (ie, within 72 hours prior to index procedure) and has elevated enzymes at time of index procedure as follows.

  * Patients are excluded if any of the following criteria are met at time of the index procedure.

    * If creatine kinase-myoglobin band (CK-MB) >2× upper limit of normal (ULN), the patient is excluded regardless of CK Total.
    * If CK-MB is 1-2× ULN, the patient is excluded if the CK Total is >2× ULN.
  * If CK Total/CK MB are not used and Troponin is, patients are excluded if the following criterion is met at time of index procedure.

    * Troponin >1× ULN with at least one of the following.
  * Patient has ischemic symptoms and ECG changes indicative of ongoing ischemia (eg, >1 mm ST segment elevation or depression in consecutive leads or new left bundle branch block [LBBB]);
  * Development of pathological Q waves in the ECG; or
  * Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.

Note: For patients with unstable angina or patients who have had a recent MI, CK Total/CK MB (or Troponin if CK Total/CK MB are not used) must be documented prior to enrolling/randomizing the patient.

* Patient has received an organ transplant or is on a waiting list for an organ transplant
* Patient is receiving or scheduled to receive chemotherapy within 30 days before or after index procedure
* Patient is receiving oral or intravenous immunosuppressive therapy (ie, inhaled steroids are not excluded) or has known life-limiting immunosuppressive or autoimmune disease (eg, human immunodeficiency virus, systemic lupus erythematosus, but not including diabetes mellitus)
* Patient is receiving chronic (>=72 hours) anticoagulation therapy (eg, heparin, coumadin) for indications other than acute coronary syndrome
* Patient has platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* Patient has white blood cell (WBC) count <3,000 cells/mm3
* Patient has documented or suspected liver disease, including laboratory evidence of hepatitis
* Patient is on dialysis or has known renal insufficiency (ie, estimated creatinine clearance <50 ml/min by the Cockcroft Gault formula, or [(140-age)*lean body weight (in kg)]/[plasma creatinine (mg/dl)*72])
* Patient has history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Patient has had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within past 6 months, or has any permanent neurologic defect that may cause non-compliance with the protocol
* Target vessel(s) or side branch has been treated with any type of PCI (eg, balloon angioplasty, stent, cutting balloon, atherectomy) within 12 months prior to index procedure
* Target vessel(s) has been treated within 10 mm proximal or distal to target lesion (by visual estimate) with any type of PCI (eg, balloon angioplasty, stent, cutting balloon, atherectomy) at any time prior to index procedure
* Non-target vessel or side branch has been treated with any type of PCI (eg, balloon angioplasty, stent, cutting balloon, atherectomy) within 24 hours prior to index procedure
* Planned or actual target vessel(s) treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon, or transluminal extraction catheter immediately prior to stent placement
* Planned PCI or CABG after index procedure
* Patient previously treated at any time with coronary intravascular brachytherapy
* Patient has a known allergy to the study stent system or protocol-required concomitant medications (eg, stainless steel, platinum, cobalt, chromium, nickel, tungsten, acrylic, fluoropolymers, everolimus, thienopyridines, aspirin, contrast) that cannot be adequately premedicated
* Patient has active peptic ulcer or active gastrointestinal (GI) bleeding
* Patient has one of the following.

  * Other serious medical illness (eg, cancer, congestive heart failure) that may reduce life expectancy to less than 24 months
  * Current problems with substance abuse (eg, alcohol, cocaine, heroin, etc.)
  * Planned procedure that may cause non-compliance with protocol or confound data interpretation
* Patient is participating in another investigational drug or device clinical trial that has not reached its primary endpoint
* Patient intends to participate in another investigational drug or device clinical trial within 12 months after index procedure
* Patient with known intention to procreate within 12 months after index procedure (Women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure.)
* Patient is a woman who is pregnant or nursing (A pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)
* Patient has more than 2 target lesions, or more than 1 target lesion and 1 non-target lesion, which will be treated during the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Maurer, MPH, Study Director — Boston Scientific Corporation
Locations (23):
- United States (14):
  - Bakersfield Memorial Hospital, Bakersfield, California
  - Mediquest Research at Munroe Regional Medical Center, Ocala, Florida
  - Florida Hospital, Orlando, Florida
  - St. John's Hospital, Springfield, Illinois
  - Jewish Hospital & St. Mary's Healthcare, Louisville, Kentucky
  - Northern Michigan Hospital, Petoskey, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Moses H. Cone Memorial Hospital/LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Ohio Health Research and Innovation Institute, Columbus, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - TexSAn Heart Hospital, San Antonio, Texas
- Australia (2):
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Monash Medical Centre, Clayton
- Belgium (2):
  - Ziekenhuis Oost Limburg, Genk
  - UZ Gasthuisberg, Leuven
- France (2):
  - Centre Hôpital Universitaire Rangueil, Toulouse, Cedex 9
  - Clinique Pasteur, Toulouse
- Japan (2):
  - Shonan Kamakura General Hospital, Kamakura-shi, Kanagawa
  - Sakurabashi Watanabe Hospital, Osaka, Osaka
- North Shore Hospital, Takapuna, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html).

REFERENCES:
- [Derived] Kelly CR, Teirstein PS, Meredith IT, Farah B, Dubois CL, Feldman RL, Dens J, Hagiwara N, Rabinowitz A, Carrie D, Pompili V, Bouchard A, Saito S, Allocco DJ, Dawkins KD, Stone GW. Long-Term Safety and Efficacy of Platinum Chromium Everolimus-Eluting Stents in Coronary Artery Disease: 5-Year Results From the PLATINUM Trial. JACC Cardiovasc Interv. 2017 Dec 11;10(23):2392-2400. doi: 10.1016/j.jcin.2017.06.070. PMID 29217001
- [Derived] Teirstein PS, Meredith IT, Feldman RL, Rabinowitz AC, Cannon LA, Lee TC, Dens J, Dubois CL, Mooney MR, Pompili VJ, Saito S, Allocco DJ, Dawkins KD, Stone GW. Two-year safety and effectiveness of the platinum chromium everolimus-eluting stent for the treatment of small vessels and longer lesions. Catheter Cardiovasc Interv. 2015 Feb 1;85(2):207-15. doi: 10.1002/ccd.25565. Epub 2014 Jul 4. PMID 24905795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of 94 patients was planned and 94 patients were enrolled at 23 sites in Australia, Belgium, France, Japan, New Zealand, and the United States from February 9, 2009 to December 10, 2009.
Period: Overall Study
Arm/Group | PROMUS Element
Started | 94
Completed | 86
Not Completed | 8
Not completed — Death | 4
Not completed — Withdrawal by Subject | 1
Not completed — Missed 12-month visit | 3

BASELINE CHARACTERISTICS:
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.33 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 68
Race/Ethnicity, Customized [Number; unit: Participant] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participant
    Hispanic or Latino | 7
    Caucasian | 80
    Asian | 4
    Black of African heritage | 4
Region of Enrollment [Number; unit: participants]
  France | 6
  United States | 75
  Belgium | 5
  Australia | 4
  Japan | 3
  New Zealand | 1
Cardiac History [Number; unit: Participant] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participant
    Previous Percutaneous Coronary Intervention (PCI) | 41
    Previous Coronary Artery Bypass Graft (CABG) | 13
    Previous Myocardial Infarction (MI) | 28
    Congestive Heart Failure | 9
    Stable Angina | 50
    Unstable Angina | 23
    Silent Ischemia | 21
Cardiac History: Ejection Fraction [Mean (Standard Deviation); unit: ejection fraction percent] | 58.07 (10.00)
Cardiac Risk Factors [Number; unit: participants] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    Smoking, Ever | 59
    Medically Treated Diabetes | 40
    Hyperlipidemia Requiring Medication | 77
    Hypertension Requiring Medication | 75
    Family History of Coronary Artery Disease | 57
Comorbidities [Number; unit: participants] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    History of Peripheral Vascular Disease | 13
    History of Transient Ischemic Attack | 5
    History of Cerebrovascular Accident | 3
    History of Renal Disease | 2
    History of Gastrointestinal Bleeding | 1
Lesion Characteristic: Target Lesion Vessel [Number; unit: lesions]
  Left Anterior Descending Artery | 32
  Left Circumflex Artery | 41
  Right Coronary Artery | 21
Lesion Characteristic: Lesion Location [Number; unit: Lesions]
  Ostial | 2
  Proximal | 40
  Mid | 37
  Distal | 15
Lesion Characteristics [Mean (Standard Deviation); unit: millimeters]
  Reference Vessel Diameter | 2.04 (0.26)
  Minimum Lumen Diameter | 0.51 (0.21)
  Lesion Length | 14.15 (7.03)
Lesion Characteristic: Percent Diameter Stenosis [Mean (Standard Deviation); unit: percent] | 75.10 (9.50)
Lesion Characteristics [Number; unit: lesions] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  lesions
    Eccentric Lesion | 66
    > 45 Degree Bend | 21
    > 90 Degree Bend | 3
    Tortuosity, any | 5
    Calcification, any | 23
    Total Occlusion | 0
    Bifurcation | 6
Lesion Characteristics: American College of Cardiology (ACC)/American Heart Association (AHA) Class [Number; unit: lesions] — Type A lesions: minimally complex, readily accessible, non-angulated, smooth contour, little to no calcification, less than totally occlusive, not ostial in location, no major side branch involvement, and an absence of thrombus.
  Type B lesions: moderately complex, eccentric, moderate tortuosity and angulation, moderate or heavy calcification, total occlusion < 3 months old, ostial in location, with presence of thrombus.
  Type C lesions: severely complex, diffuse, excessive tortuosity and angulation, total occlusions > 3 months old, degenerated vein grafts and friable lesions.
  lesions
    Type A | 8
    Type B1 | 21
    Type B2 | 41
    Type C | 24
Lesion Characteristic - Pre-Procedure Thrombolysis In Myocardial Infarction (TIMI) Flow [Number; unit: participants] — TIMI 0 - No perfusion; TIMI 1 - Penetration with minimal perfusion; TIMI 2 - Partial perfusion; TIMI 3 - Complete perfusion
  participants
    TIMI 0 | 0
    TIMI 1 | 0
    TIMI 2 | 6
    TIMI 3 | 88

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Failure (TLF)
Description: Defined as any ischemia-driven revascularization of the target lesion, myocardial infarction (Q-wave and non-Q-wave) related to the target vessel, or cardiac death related to the target vessel. The primary analysis set for the non-inferiority testing of the primary endpoint is the per-protocol analysis set. All randomized participants who received their assigned treatment are included in the per-protocol analysis set.
Time Frame: 12 Months
Population: The primary analysis set for comparison of the primary endpoint, 12-month TLF, to the predefined performance goal of 21.1% (based on historical TAXUS Express results) is the per-protocol analysis set. All enrolled participants who received a PROMUS Element stent are included in the per-protocol analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 84
percentage of participants | 2.4
Statistical Analysis 1: Comparison: PROMUS Element; A one-group exact binomial test was used to test the hypothesis that the primary endpoint rate in the PROMUS Element cohort is less than the predefined performance goal of 21.1%; Test type: Superiority or Other; p < 0.0001, One-group exact binomial test; Percent Target Lesion Failure = 2.4, 95% CI 1-sided [upper limit 7.3]

2. Secondary Outcome: Target Lesion Failure (TLF)
Description: Defined as any ischemia-driven revascularization of the target lesion, myocardial infarction (Q-wave and non-Q-wave) related to the target vessel, or cardiac death related to the target vessel.
Time Frame: 6 Months
Population: Analysis was intention to treat; all patients in the study underwent clinical follow up to provide the information needed for this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 93
percentage of participants | 3.2

3. Secondary Outcome: Target Lesion Failure (TLF)
Description: as for outcome 2
Time Frame: 30 Days
Population: Analysis was intention to treat; all participants underwent clinical follow-up to provide the information needed for this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants | 0.0

4. Secondary Outcome: Target Vessel Failure (TVF)
Description: Target vessel failure (TVF) is defined as any ischemia-driven revascularization of the target vessel, myocardial infarction (MI;Q-wave and non-Q-wave) related to the target vessel or death related to the target vessel. For the purposes of this protocol, if it cannot be determined with certainty whether the MI or death was related to the target vessel, it will be considered a TVF.
Time Frame: 12 Months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 89
percentage of participants | 6.7

5. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 4
Time Frame: 6 Months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 93
percentage of participants | 4.3

6. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 4
Time Frame: 30 Days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants | 0.0

7. Secondary Outcome: Myocardial Infarction (MI) Related to the Target Vessel
Description: New Q-waves in ≥2 leads lasting ≥0.04 sec with creatine kinase myoglobin band(CK-MB) or troponin >upper limit of normal(ULN); if no new Q-waves total CK levels >3×ULN (peri-percutaneous coronary intervention [PCI]) or >2×ULN (spontaneous) with elevated CK-MB or troponin >3×ULN (peri-PCI) or >2×ULN (spontaneous) plus ≥one of the following: ECG changes indicating new ischemia (new ST-T changes, left bundle branch block), imaging evidence of new loss of viable myocardium, new regional wall motion abnormality. Similar for MI diagnosis post coronary artery bypass graft with CK-MB or troponin >5×ULN
Time Frame: 12 Months
Population: as for outcome 2
Measure: Number; unit: percentage of participants with MI
Arm/Group | PROMUS Element
Number analyzed (Participants) | 90
percentage of participants with MI | 0.0

8. Secondary Outcome: Myocardial Infarction (MI) Related to the Target Vessel
Description: as for outcome 7
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants with MI
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants with MI | 0.0

9. Secondary Outcome: Myocardial Infarction (MI) Related to the Target Vessel
Description: as for outcome 7
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants with MI
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants with MI | 0.0

10. Secondary Outcome: All Cause Mortality
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 90
percentage of participants | 4.4

11. Secondary Outcome: All Cause Mortality
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants | 2.1

12. Secondary Outcome: All Cause Mortality
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants | 0.0

13. Secondary Outcome: Cardiac Death Related to the Target Vessel
Description: Defined as death due to any of the following: acute myocardial infarction (MI); cardiac perforation/pericardial tamponade; arrhythmia or conduction abnormality; cerebrovascular accident (CVA) through hospital discharge or CVA suspected of being related to the procedure; complication of the procedure including bleeding, vascular repair, transfusion reaction, or bypass surgery or any death in which a cardiac cause cannot be excluded; see definition of MI above.
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 90
percentage of participants | 3.3

14. Secondary Outcome: Cardiac Death Related to the Target Vessel
Description: Cardiac death is defined as death due to any of the following: acute myocardial infarction (MI); cardiac perforation/pericardial tamponade; arrhythmia or conduction abnormality; cerebrovascular accident (CVA) through hospital discharge or CVA suspected of being related to the procedure; complication of the procedure including bleeding, vascular repair, transfusion reaction, or bypass surgery or any death in which a cardiac cause cannot be excluded; see definition of MI above
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants | 1.1

15. Secondary Outcome: Cardiac Death Related to the Target Vessel
Description: as for outcome 14
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants | 0.0

16. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: Defined as any ischemia-driven repeat percutaneous intervention to improve blood flow of the successfully treated target lesion or bypass surgery of the target vessel with a graft distally to the successfully treated target lesion.
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants with TLR
Arm/Group | PROMUS Element
Number analyzed (Participants) | 90
percentage of participants with TLR | 2.2

17. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: as for outcome 16
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants with TLR
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants with TLR | 2.1

18. Secondary Outcome: Target Lesion Revascularization TLR)
Description: as for outcome 16
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants with TLR
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants with TLR | 0.0

19. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: Defined as any ischemia-driven repeat percutaneous intervention to improve blood flow, or bypass surgery of not previously existing lesions with diameter stenosis ≥50% by quantitative coronary angiography in the target vessel, including the target lesion.
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants with TVR
Arm/Group | PROMUS Element
Number analyzed (Participants) | 90
percentage of participants with TVR | 3.3

20. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: as for outcome 19
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants with TVR
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants with TVR | 3.2

21. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: Any ischemia-driven repeat percutaneous intervention to improve blood flow, or bypass surgery of not previously existing lesions with diameter stenosis ≥50% by quantitative coronary angiography in the target vessel, including the target lesion.
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants with TVR
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants with TVR | 0.0

22. Secondary Outcome: Definite + Probable Stent Thrombosis (ST) Rate Based on Academic Research Consortium (ARC)Definition
Description: DEFINITE ST: acute coronary syndrome and angiographic or pathologic evidence of stent thrombosis; PROBABLE ST: unexplained death within 30 days or target-vessel infarction without angiographic information ARC ST is reported as a cumulative value at different time points and within the different separate time points. Time 0 is the time point after the guide catheter has been removed. Acute ST: 0-24 hours after stent implantation; Subacute ST: >24 hours to 30 days post; late ST: >30 days to 1 year post; Very late ST: >1 year post; NOTE: Acute/subacute can be replaced by early ST (0-30 days)
Time Frame: 24 hours
Population: as for outcome 2
Measure: Number; unit: percentage of participants with ST
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants with ST | 0.0

23. Secondary Outcome: Definite + Probable Stent Thrombosis (ST) Rate Based on Academic Research Consortium (ARC) Definition
Description: as for outcome 22
Time Frame: >24 hr-30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants with ST
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants with ST | 0

24. Secondary Outcome: Definite + Probable Stent Thrombosis (ST) Rate Based on Academic Research Consortium (ARC) Definition
Description: as for outcome 22
Time Frame: >30 days-1 year
Population: as for outcome 2
Measure: Number; unit: percentage of participants with ST
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants with ST | 0.0

25. Secondary Outcome: Acute Technical Success
Description: Defined as successful delivery and deployment of the study stent to the target vessel, without balloon rupture or stent embolization; expressed per stent
Time Frame: During the index procedure (minutes)
Population: Analysis was intention to treat
Measure: Number; unit: percentage of stents
Units Other Than Participants: stents
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
Number analyzed (stents) | 95
percentage of stents | 96.8

26. Secondary Outcome: Clinical Procedural Success
Description: Defined as mean lesion diameter stenosis <30% with visually assessed TIMI 3 flow and without the occurrence of in-hospital MI, TVR, or cardiac death.
Time Frame: Duration of Hospital Stay (average 1-2 days)
Population: Analysis was intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 94
percentage of participants | 96.8

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | PROMUS Element
Serious Adverse Events (participants affected / at risk) | 27/94
Other Adverse Events (participants affected / at risk) | 31/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMUS Element (N=94)
Angina pectoris (Cardiac disorders) | 7 (11)
Myocardial infarction (Cardiac disorders) | 5 (6)
Angina unstable (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (4)
Death (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Arteriosclerosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gunshot wound (Injury, poisoning and procedural complications) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMUS Element (N=94)
Adverse drug reaction (General disorders) | 9 (9)
Non-cardiac chest pain (General disorders) | 7 (7)
Catheter site haematoma (General disorders) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Angina pectoris (Cardiac disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) shall have the right to publish the results, provided that before publishing, the PI shall submit copies of any proposed publication or presentation to the Sponsor for review at least 45 days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any confidential information or other proprietary information of Sponsor from the proposed publication or presentation.